CLINICAL TRIAL: NCT03773861
Title: Determining a Threshold for the Clinical and Cost-effectiveness of Group Size During Basic Life Support Courses
Brief Title: Group Size in Basic Life Support (BLS) Courses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Req- 2017- 00577
Record Dates: First submitted 2018-11-28; First posted 2018-12-12 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Educational Problems; Resuscitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants (Other): Active BLS- Instructors at the Bern Simulation and CPR- Center (BeSiC), at the Bern University Hospital, Bern, Switzerland. Participants have to oversee a BLS instructional session, where standardized errors are performed by trained volunteers.
  Interventions: Other: errors made in one BLS session

INTERVENTIONS:
Other: errors made in one BLS session — BLS instructors have to oversee a standardized BLS training session, where standardized errors are made by trained volunteers.

SUMMARY:
Basic Life Support (BLS) is important for outcome in cardiac arrest.Therefore, it is crucial to improve the quality of education in resuscitation training. Better training will eventually lead to more effective CPR skills in course participants. BLS courses in both international resuscitation associations (European Resuscitation Council and American Heart Association are typically taught in small groups of 6 participants. In reality group sizes of up to 10 participants are used, because these courses are highly demanded and cost intensive. There is no evidence for the effective group size to be clinical and cost effective. Therefore the investigators perform this prospective study to determine the maximum number of participants an instructor can oversee without missing more than 20% of errors made during an instructional BLS session.

ELIGIBILITY:
Inclusion Criteria:

* Active BLS- Instructors at the Bern Simulation and CPR-Center (BeSiC), at the Bern University Hospital, Bern, Switzerland

Exclusion Criteria:

* Decline to participate

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2018-12-10 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
The threshold of number of course participants in a BLS educational session | BLS educational session 10 minutes
  How many volunteers can be overseen by one instructor who still is able to correctly identify and correct serious BLS errors of all course participants.

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Nabecker, M.D., Principal Investigator — University Hospital Bern, Bern, Switzerland
Locations (1):
- University Hospital Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Perkins GD, Handley AJ, Koster RW, Castren M, Smyth MA, Olasveengen T, Monsieurs KG, Raffay V, Grasner JT, Wenzel V, Ristagno G, Soar J; Adult basic life support and automated external defibrillation section Collaborators. European Resuscitation Council Guidelines for Resuscitation 2015: Section 2. Adult basic life support and automated external defibrillation. Resuscitation. 2015 Oct;95:81-99. doi: 10.1016/j.resuscitation.2015.07.015. Epub 2015 Oct 15. No abstract available. PMID 26477420
- [Background] Beck S, Issleib M, Daubmann A, Zollner C. Peer education for BLS-training in schools? Results of a randomized-controlled, noninferiority trial. Resuscitation. 2015 Sep;94:85-90. doi: 10.1016/j.resuscitation.2015.06.026. Epub 2015 Jul 14. PMID 26184655
- [Background] Cendan JC, Silver M, Ben-David K. Changing the student clerkship from traditional lectures to small group case-based sessions benefits the student and the faculty. J Surg Educ. 2011 Mar-Apr;68(2):117-20. doi: 10.1016/j.jsurg.2010.09.011. PMID 21338967
- [Background] Chamberlain DA, Hazinski MF; European Resuscitation Council; American Heart Association; Heart and Stroke Foundation of Canada; Resuscitation Council of Southern Africa; Australia and New Zealand Resuscitation Council; Consejo Latino-Americano de Resusucitacion. Education in resuscitation: an ILCOR symposium: Utstein Abbey: Stavanger, Norway: June 22-24, 2001. Circulation. 2003 Nov 18;108(20):2575-94. doi: 10.1161/01.CIR.0000099898.11954.3B. No abstract available. PMID 14623795